CLINICAL TRIAL: NCT04272190
Title: Effect of Different Treatments on the Prognosis of Early Cervical Cancer: A Multicenter, Prospective, Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Chen Chunlin, Director of Department of Obstetrics and Gynecology, Southern Medical University, China
Other Study IDs: NFEC-2019-105
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Preoperative treatment; Surgical approach; Hysterectomy type; Radiochemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical routine treatments — The cohort stratified by four factors: preoperative treatment (not received, neoadjuvant chemotherapy, preoperative radiotherapy); surgical approach (laparoscopic, abdominal, vaginal, robotic); hysterectomy types (type A, type B, type C1, type C2), primary treatment (Radical hysterectomy + pelvic lymph node dissectionp; radiochemotherapy)

SUMMARY:
To observe the effects of different treatments on the oncological outcome and complications of early cervical cancer (2018 FIGO stage IA1 with lymphovascular space invasion and IA2-IIA2 cervical cancer). This study prospectively collecting enrolled cervical cancer patients clinical data and outcome from June 2020 to June 2025. (Classification factors: preoperative neoadjuvant treatment , surgical approach, type of hysterectomy, whether to receive radiochemotherapy) . This study is an observational study, and segmented analysis according to different treatment methods.

DETAILED DESCRIPTION:
Objectives: To observe the effects of different treatments on the oncological outcome and complications of early cervical cancer (2018 FIGO stage IA1 with lymphovascular space invasion and IA2-IIA2 cervical cancer).

Study Design: We obtained the demographic, clinical, treatment hospital and complication data of patients with cervical cancer undergoing radical hysterectomy from 2004 to 2015 at 37 hospitals. The patients were assigned into groups. Classification factors: preoperative neoadjuvant treatment (not received, neoadjuvant chemotherapy, preoperative radiotherapy) , surgical approach (abdomincal, laparoscopic, vaginal, robotic surgery), type of hysterectomy (type B, type C1, type C2), primary treatment (radiochemotherapy or surgery).

laparoscopic and abdominal surgery groups. The differences in the survival, complication rates, quality of life, and cost were analyzed using univariate and multivariable logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary adenocarcinoma, squamous cell carcinoma, adenosquamous carcinoma, or other histological types carcinoma of the uterine cervix.
2. Patients with Histologically confirmed stage IA1 (with lymph vascular invasion), FIGO 2018 stage IA2 to IIA2.
3. Underwent radical hysterectomy or radiochemotherapy.
4. ECOG Performance Status of 0 or 1.

Exclusion Criteria:

1. Life expectancy is less than 6 months
2. No prior malignancy
3. ECOG Performance Status of 2 to 5.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 60 months from primary treatment
  Overall survival was defined as the period from initial treatment until cervical cancer related death.
disease-free survival (DFS) | 60 months from primary treatment
  Tumor-free survival was defined as the period from initial treatment until the recurrence or the date of last follow-up.

SECONDARY OUTCOMES:
Patterns of recurrence | 60 months from primary treatment
  date and localization of 1st recurrence as confirmed histologically
Costs of treatment | 60 months from primary treatment
Costs of readmission | 60 months from primary treatment
Quality of life Questionnaires | 60 months from primary treatment
  The European O-rganization for Reasearch and Treatment of Cance QLQ-30 Questionnaires to measure quality of life for any kind cancer patient. The Europe Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Cervical Cancer Module is a supplementary questionnaire for evaluating the quality of life of patients with cervical cancer.
The morbidity of sexual dysfunction | 60 months from primary treatment
  Female Sexual Function Index (FSFI)
Intra-operative, peri-operative, post-operative and long term treatment related morbidity | 60 months from primary treatment
  Complications of all the patients

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chunlin, PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided